CLINICAL TRIAL: NCT01795391
Title: Comparison Between Two New Generation Dressings in the Prevention of Intravascular Catheter Related Complications in Intensive Care Units
Brief Title: Comparison of Two New Generations Dressings in Intensive Care Unit
Acronym: Advanced
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: ADVANCED
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Catheter Related Complications
Keywords: Prevention; Dressings; Catheters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Tegaderm HP: Patients whose intravasculare devices dressings are made exclusevely with Tegaderm HP dressings.
- Advanced: Patients whose intravasculare devices dressings are made exclusevely with Advanced dressings

SUMMARY:
Intravascular devices in intensive care units are often associated to complications. The investigators estimate that 23.5% of catheters placed and used in intensive care are subject to at least one complication; the goal is to demonstrate the effectiveness of the new Tegaderm ™ IV Advanced dressings to achieve a decrease of 35% in the number of complications associated with intravascular catheters in intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years with a central venous catheter, an arterial catheter, a hemodialysis catheter, a Swan Ganz catheter or a peripheral catheter inserted in the ICU or within the 24 before their arrival at the ICU in another ICU setting.
* Patients benefiting from the social security protection.

Exclusion Criteria:

* Patients under 18 years of age,
* Patients having known allergy or sensitivity to adhesive dressing materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalised in the Medical ICU and requiring an intravascular device during hospitalisation (peripheral or central)
Sampling Method: Probability Sample
Enrollment: 685 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of catheters presenting any kind of complications. | From the insertion of the catheter to its removal, an average time frame thant can go up to 4 weeks.

SECONDARY OUTCOMES:
Number of infections related to poor adherent dressings. | From the insertion of the catheter to its removal, an average time frame thant can go up to 4 weeks.

OTHER OUTCOMES:
Number of participants presenting allergic adverse events. | From the insertion of the catheter to its removal, an average time frame thant can go up to 4 weeks.
Cost of each dressing type strategy. | From the insertion of the catheter to its removal, an average time frame thant can go up to 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Grenoble, Medical Intensive Care Unit, Grenoble, Isère, France